CLINICAL TRIAL: NCT04904406
Title: Changes in Weight and Body Composition After Switch to Dolutegravir/Lamivudine Compared to Continued Dolutegravir/Abacavir/Lamivudine for Virologically Suppressed HIV Infection: A Randomized Open-label Superiority Trial: AVERTAS-1
Brief Title: Changes in Weight, Body Composition and Cardiac Risk After Discontinuing Abacavir Treatment in HIV-infected Individuals
Acronym: AVERTAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Benfield (Other)
Responsible Party: Sponsor-Investigator, Thomas Benfield, MD, DMsc, professor,, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-20011433
Record Dates: First submitted 2020-10-09; First posted 2021-05-27 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Hiv; HIV Infections; HIV Cardiomyopathy; Weight Change, Body; HIV Lipodystrophy; Cardiovascular Diseases
Keywords: HIV; Weight changes; Antiretroviral Therapy; Cardiovascular disease; Antiretroviral therapy side effects; Antiretroviral two-drug regimen; HIV metabolism; HIV diabetes
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Body Weight Changes; Cardiovascular Diseases | interventions — dolutegravir; Lamivudine; abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Intervention Model Description: A randomized controlled open-label superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dolutegravir/lamivudine (Experimental): 50 mg dolutegravir and 300 mg lamivudine (co-formulated) once daily for 48 weeks
  Interventions: Drug: Dolutegravir / Lamivudine Oral Tablet
- dolutegravir/abacavir/lamivudine (No Intervention): 50 mg dolutegravir, 600 mg abacavir and 300 mg lamivudine (co-formulated) once daily for 48 weeks

INTERVENTIONS:
Drug: Dolutegravir / Lamivudine Oral Tablet — Discontinuing abacavir by switching from three-drug regimen with dolutegravir/abacavir/lamivudine to two-drug regimen with dolutegravir/lamivudine
  Other Names: Dolutegravir/abacavir/lamivudine
  Arms: dolutegravir/lamivudine

SUMMARY:
Randomized controlled parallel open-label study in people living with HIV and at least 6 month of treatment with dolutegravir/abacavir/lamivudine prior to inclusion.

Participants (n=95) are randomized to continue 3 drug-regimen dolutegravir/abacavir/lamivudine (control) or switch to two-drug regimen with dolutegravir/lamivudine (intervention). Follow-up is 48 weeks. Data is collected at baseline and week 48. Primary outcome is changes in weight from baseline of more than 2 kg. Secondary outcomes are changes in cardiac risk, composition and calcification of the heart tissue, and changes in body composition and metabolism, inflammation and coagulation. A MRI substudy is applied to focus on the cardiac adverse effects of abacavir.

DETAILED DESCRIPTION:
In the MRI sub study 40 patients from the main study (20 from each group) are included. A cardiac MRI are performed at baseline and week 48 to evaluate cardiac effects of abacavir.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Diagnosed HIV
* At least 6 months of ongoing treatment with dolutegravir/ abacavir/lamivudine
* Plasma viral load (HIV-RNA) < 50 copies/ml at inclusion

For women of childbearing potential:

* Negative pregnancy test
* Willingness to use contraceptive (consistent with local regulations) during study period

Exclusion Criteria:

* Pre-existing viral resistance mutations to lamivudine or to dolutegravir
* Presence of hepatitis B antigen (HBsAg) or Hepatitis B virus DNA (HBV DNA)
* Cancer within past 5 years
* Diabetes, cardiovascular disease or other chronic illness considered stable as assessed by the treating physician

For women of childbearing potential:

* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in body weight of ≥2 kg | 48 weeks
  Fasting body weight

SECONDARY OUTCOMES:
Virological control | 48 weeks
  HIV-RNA <50 copies/ml
Changes in self-rated health | 48 weeks
  12-item Short Form Health Survey (SF-12). Scores from 0 (worse) to 100 (best).
Change in metabolism | 48 weeks
  Impaired insulin resistance and/or β-cell function determined by changes in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Changes in cardiac risk | 48 weeks
  D:A:D CVD risk score: Five and ten years predicted cardio vascular disease risk (percent)
Changes in carotid artery intima-media thickness (cIMT) | 48 weeks
  Measured by ultrasound.
Changes in Coronary artery calcium score (CACS) | 48 weeks
  Measures by CT-scan. Scores from 0 and with no upper limit. The higher score, the worse calcification/plaque level and higher CVD risk.
Changes in cardiac blood markers | 48 weeks
  Changes in N-terminal pro-B-type natriuretic peptide (Pro-BNP)
Changes in bloodpressure | 48 weeks
  Systolic and diastolic blood pressure (mmHg)
Changes in fat distribution VAT/SAT | 48 weeks
  Measured by CT-scan
  • Visceral adipose tissue (VAT) and subcutaneous adipose tissue (SAT) determined by abdominal CT.
Changes in liver stiffness | 48 weeks
  Measured by CT-scan and liver elastography
Changes in liver fat infiltration | 48 weeks
  Measured by CT-scan and liver elastography
Changes in fat distribution in trunk, limb and extremities | 48 weeks
  Measured by dual energy xray absorptiometry (DEXA)
Changes in inflammation | 48 weeks
  High-sensitive C-reactive protein
Changes in interleukins | 48 weeks
  Interleukin 1- and interleukin 6
Changes in endothelial function | 48 weeks
  Vascular cell adhesion molecule 1 and intercellular adhesion molecule 1
Changes in soluble P-selectin | 48 weeks
  soluble P-selectin
Changes in soluble glycoprotein VI | 48 weeks
  soluble glycoprotein VI
Changes in d-dimer | 48 weeks
  D-dimer
Changes in coagulation | 48 weeks
  Factor 2, 7 and 10 (extrinsic pathway)
Changes in fibrinogen | 48 weeks
  Fibrinogen
Changes in blood Hemoglobin | 48 weeks
  Hemoglobin
Changes in blood platelets | 48 weeks
  Platelets
Changes in plasma creatinine | 48 weeks
  Creatinine
Changes in plasma urea | 48 weeks
  Urea
Changes in plasma sodium | 48 weeks
  Sodium
Changes in plasma potassium | 48 weeks
  Potassium
Changes in plasma bilirubin | 48 weeks
  Bilirubin
Changes in plasma alanine | 48 weeks
  Alanine
Changes in plasma aminotransferase | 48 weeks
  Aminotransferase
Cardiovascular risk | 48 weeks
  Framingham risk score: Estimated 10 years risk of cardiovascular disease (percent)
Cardiac biomarkers | 48 weeks
  Changes in Troponin T (TnT)

OTHER OUTCOMES:
Cardiac MRI substudy primary outcome (composite) ECV | 48 weeks
  Cardiac MRI applied on 40 patients to evaluate:
  Decrease in extracellular myocardial volume (ECV) from baseline to week 48
Cardiac MRI substudy primary outcome (composite) atrial volume | 48 weeks
  Cardiac MRI applied on 40 patients to evaluate:
  Decrease in left atrial volume from baseline to week 48
Cardiac MRI substudy primary outcome (composite) diastolic function | 48 weeks
  Cardiac MRI applied on 40 patients to evaluate:
  Improvement in diastolic function from baseline to week 48
Cardiac MRI substudy primary outcome (composite) myocardial mass | 48 weeks
  Cardiac MRI applied on 40 patients to evaluate:
  Reduction in myocardial mass from baseline to week 48
Cardiac MRI substudy secondary outcome ejection fraction (EF) | 48 weeks
  Cardiac MRI applied on 40 patients to evaluate:
  Secondary outcomes
  Changes in:
  • Ejection fraction (EF)
Cardiac MRI substudy secondary outcome perfusion | 48 weeks
  Cardiac MRI applied on 40 patients to evaluate:
  Secondary outcomes
  Changes in:
  • Perfusion
Cardiac MRI substudy secondary outcome edema/inflammation | 48 weeks
  Cardiac MRI applied on 40 patients to evaluate:
  Secondary outcomes
  Changes in:
  • Edema/inflammation
Cardiac MRI substudy secondary outcome fibrosis | 48 weeks
  Cardiac MRI applied on 40 patients to evaluate:
  Secondary outcomes
  Changes in:
  • Fibrosis
Cardiac MRI substudy secondary outcome lipid | 48 weeks
  Cardiac MRI applied on 40 patients to evaluate:
  Secondary outcomes
  Changes in:
  • Lipid-water profile Measured by MR spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Benfield, MD, DMSc, Principal Investigator — Department of Infectious diseases, Hvidovre Hospital, Denmark
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Copenhagen University Hospital, Amager Hvidovre, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belloso WH, Orellana LC, Grinsztejn B, Madero JS, La Rosa A, Veloso VG, Sanchez J, Ismerio Moreira R, Crabtree-Ramirez B, Garcia Messina O, Lasala MB, Peinado J, Losso MH. Analysis of serious non-AIDS events among HIV-infected adults at Latin American sites. HIV Med. 2010 Oct 1;11(9):554-64. doi: 10.1111/j.1468-1293.2010.00824.x. Epub 2010 Mar 21. PMID 20345879
- [Background] Smith CJ, Ryom L, Weber R, Morlat P, Pradier C, Reiss P, Kowalska JD, de Wit S, Law M, el Sadr W, Kirk O, Friis-Moller N, Monforte Ad, Phillips AN, Sabin CA, Lundgren JD; D:A:D Study Group. Trends in underlying causes of death in people with HIV from 1999 to 2011 (D:A:D): a multicohort collaboration. Lancet. 2014 Jul 19;384(9939):241-8. doi: 10.1016/S0140-6736(14)60604-8. PMID 25042234
- [Background] Freiberg MS, Chang CC, Kuller LH, Skanderson M, Lowy E, Kraemer KL, Butt AA, Bidwell Goetz M, Leaf D, Oursler KA, Rimland D, Rodriguez Barradas M, Brown S, Gibert C, McGinnis K, Crothers K, Sico J, Crane H, Warner A, Gottlieb S, Gottdiener J, Tracy RP, Budoff M, Watson C, Armah KA, Doebler D, Bryant K, Justice AC. HIV infection and the risk of acute myocardial infarction. JAMA Intern Med. 2013 Apr 22;173(8):614-22. doi: 10.1001/jamainternmed.2013.3728. PMID 23459863
- [Background] Sabin CA, Reiss P, Ryom L, Phillips AN, Weber R, Law M, Fontas E, Mocroft A, de Wit S, Smith C, Dabis F, d'Arminio Monforte A, El-Sadr W, Lundgren JD; D:A:D Study Group. Is there continued evidence for an association between abacavir usage and myocardial infarction risk in individuals with HIV? A cohort collaboration. BMC Med. 2016 Mar 31;14:61. doi: 10.1186/s12916-016-0588-4. PMID 27036962
- [Background] Worm SW, Sabin C, Weber R, Reiss P, El-Sadr W, Dabis F, De Wit S, Law M, Monforte AD, Friis-Moller N, Kirk O, Fontas E, Weller I, Phillips A, Lundgren J. Risk of myocardial infarction in patients with HIV infection exposed to specific individual antiretroviral drugs from the 3 major drug classes: the data collection on adverse events of anti-HIV drugs (D:A:D) study. J Infect Dis. 2010 Feb 1;201(3):318-30. doi: 10.1086/649897. PMID 20039804
- [Background] D:A:D Study Group; Sabin CA, Worm SW, Weber R, Reiss P, El-Sadr W, Dabis F, De Wit S, Law M, D'Arminio Monforte A, Friis-Moller N, Kirk O, Pradier C, Weller I, Phillips AN, Lundgren JD. Use of nucleoside reverse transcriptase inhibitors and risk of myocardial infarction in HIV-infected patients enrolled in the D:A:D study: a multi-cohort collaboration. Lancet. 2008 Apr 26;371(9622):1417-26. doi: 10.1016/S0140-6736(08)60423-7. Epub 2008 Apr 2. PMID 18387667
- [Background] Venter WDF, Moorhouse M, Sokhela S, Fairlie L, Mashabane N, Masenya M, Serenata C, Akpomiemie G, Qavi A, Chandiwana N, Norris S, Chersich M, Clayden P, Abrams E, Arulappan N, Vos A, McCann K, Simmons B, Hill A. Dolutegravir plus Two Different Prodrugs of Tenofovir to Treat HIV. N Engl J Med. 2019 Aug 29;381(9):803-815. doi: 10.1056/NEJMoa1902824. Epub 2019 Jul 24. PMID 31339677
- [Background] Lake JE, Wu K, Bares SH, Debroy P, Godfrey C, Koethe JR, McComsey GA, Palella FJ, Tassiopoulos K, Erlandson KM. Risk Factors for Weight Gain Following Switch to Integrase Inhibitor-Based Antiretroviral Therapy. Clin Infect Dis. 2020 Dec 3;71(9):e471-e477. doi: 10.1093/cid/ciaa177. PMID 32099991
- [Background] Hill A, Waters L, Pozniak A. Are new antiretroviral treatments increasing the risks of clinical obesity? J Virus Erad. 2019 Jan 1;5(1):41-43. doi: 10.1016/S2055-6640(20)30277-6. PMID 30800425
- [Background] Sax PE, Erlandson KM, Lake JE, Mccomsey GA, Orkin C, Esser S, Brown TT, Rockstroh JK, Wei X, Carter CC, Zhong L, Brainard DM, Melbourne K, Das M, Stellbrink HJ, Post FA, Waters L, Koethe JR. Weight Gain Following Initiation of Antiretroviral Therapy: Risk Factors in Randomized Comparative Clinical Trials. Clin Infect Dis. 2020 Sep 12;71(6):1379-1389. doi: 10.1093/cid/ciz999. PMID 31606734
- [Background] Choi AI, Vittinghoff E, Deeks SG, Weekley CC, Li Y, Shlipak MG. Cardiovascular risks associated with abacavir and tenofovir exposure in HIV-infected persons. AIDS. 2011 Jun 19;25(10):1289-98. doi: 10.1097/QAD.0b013e328347fa16. PMID 21516027
- [Background] Desai M, Joyce V, Bendavid E, Olshen RA, Hlatky M, Chow A, Holodniy M, Barnett P, Owens DK. Risk of cardiovascular events associated with current exposure to HIV antiretroviral therapies in a US veteran population. Clin Infect Dis. 2015 Aug 1;61(3):445-52. doi: 10.1093/cid/civ316. Epub 2015 Apr 22. PMID 25908684
- [Background] O'Halloran JA, Dunne E, Tinago W, Denieffe S, Kenny D, Mallon PWG. Switching from abacavir to tenofovir disoproxil fumarate is associated with rises in soluble glycoprotein VI, suggesting changes in platelet-collagen interactions. AIDS. 2018 Apr 24;32(7):861-866. doi: 10.1097/QAD.0000000000001783. PMID 29438200
- [Background] Freiberg MS, Chang CH, Skanderson M, Patterson OV, DuVall SL, Brandt CA, So-Armah KA, Vasan RS, Oursler KA, Gottdiener J, Gottlieb S, Leaf D, Rodriguez-Barradas M, Tracy RP, Gibert CL, Rimland D, Bedimo RJ, Brown ST, Goetz MB, Warner A, Crothers K, Tindle HA, Alcorn C, Bachmann JM, Justice AC, Butt AA. Association Between HIV Infection and the Risk of Heart Failure With Reduced Ejection Fraction and Preserved Ejection Fraction in the Antiretroviral Therapy Era: Results From the Veterans Aging Cohort Study. JAMA Cardiol. 2017 May 1;2(5):536-546. doi: 10.1001/jamacardio.2017.0264. PMID 28384660
- [Background] Thiara DK, Liu CY, Raman F, Mangat S, Purdy JB, Duarte HA, Schmidt N, Hur J, Sibley CT, Bluemke DA, Hadigan C. Abnormal Myocardial Function Is Related to Myocardial Steatosis and Diffuse Myocardial Fibrosis in HIV-Infected Adults. J Infect Dis. 2015 Nov 15;212(10):1544-51. doi: 10.1093/infdis/jiv274. Epub 2015 May 11. PMID 25964507
- [Background] Luetkens JA, Doerner J, Schwarze-Zander C, Wasmuth JC, Boesecke C, Sprinkart AM, Schmeel FC, Homsi R, Gieseke J, Schild HH, Rockstroh JK, Naehle CP. Cardiac Magnetic Resonance Reveals Signs of Subclinical Myocardial Inflammation in Asymptomatic HIV-Infected Patients. Circ Cardiovasc Imaging. 2016 Mar;9(3):e004091. doi: 10.1161/CIRCIMAGING.115.004091. PMID 26951603
- [Background] Ntusi N, O'Dwyer E, Dorrell L, Wainwright E, Piechnik S, Clutton G, Hancock G, Ferreira V, Cox P, Badri M, Karamitsos T, Emmanuel S, Clarke K, Neubauer S, Holloway C. HIV-1-Related Cardiovascular Disease Is Associated With Chronic Inflammation, Frequent Pericardial Effusions, and Probable Myocardial Edema. Circ Cardiovasc Imaging. 2016 Mar;9(3):e004430. doi: 10.1161/CIRCIMAGING.115.004430. PMID 26951605
- [Background] Friis-Moller N, Thiebaut R, Reiss P, Weber R, Monforte AD, De Wit S, El-Sadr W, Fontas E, Worm S, Kirk O, Phillips A, Sabin CA, Lundgren JD, Law MG; DAD study group. Predicting the risk of cardiovascular disease in HIV-infected patients: the data collection on adverse effects of anti-HIV drugs study. Eur J Cardiovasc Prev Rehabil. 2010 Oct;17(5):491-501. doi: 10.1097/HJR.0b013e328336a150. PMID 20543702
- [Background] Hsue PY, Hunt PW, Ho JE, Farah HH, Schnell A, Hoh R, Martin JN, Deeks SG, Bolger AF. Impact of HIV infection on diastolic function and left ventricular mass. Circ Heart Fail. 2010 Jan;3(1):132-9. doi: 10.1161/CIRCHEARTFAILURE.109.854943. Epub 2009 Nov 20. PMID 19933410
- [Background] Hutchins E, Wang R, Rahmani S, Nakanishi R, Haberlen S, Kingsley L, Witt MD, Palella FJ Jr, Jacobson L, Budoff MJ, Post WS. HIV Infection Is Associated with Greater Left Ventricular Mass in the Multicenter AIDS Cohort Study. AIDS Res Hum Retroviruses. 2019 Aug;35(8):755-761. doi: 10.1089/AID.2019.0014. Epub 2019 Jun 3. PMID 31044604
- [Background] Erqou S, Lodebo BT, Masri A, Altibi AM, Echouffo-Tcheugui JB, Dzudie A, Ataklte F, Choudhary G, Bloomfield GS, Wu WC, Kengne AP. Cardiac Dysfunction Among People Living With HIV: A Systematic Review and Meta-Analysis. JACC Heart Fail. 2019 Feb;7(2):98-108. doi: 10.1016/j.jchf.2018.10.006. PMID 30704613
- [Derived] Pedersen KBH, Knudsen A, Moller S, Siebner HR, Hove JD, Gerstoft J, Benfield T. Changes in weight, body composition and metabolic parameters after switch to dolutegravir/lamivudine compared with continued treatment with dolutegravir/abacavir/lamivudine for virologically suppressed HIV infection (The AVERTAS trial): a randomised, open-label, superiority trial in Copenhagen, Denmark. BMJ Open. 2023 Aug 21;13(8):e075673. doi: 10.1136/bmjopen-2023-075673. PMID 37604629